CLINICAL TRIAL: NCT04853589
Title: Effect of Hyaluronic Acid on the Therapy of Alveolar Osteitis - A Double-blind, Randomized Controlled Clinical Trial
Brief Title: Effect of Hyaluronic Acid on the Therapy of Alveolar Osteitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Danijel Domic DMD, Dental medical doctor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1049/2021
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Alveolar Osteitis
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic acid (Active Comparator): hyaluronic acid gel application
  Interventions: Device: Hyaluronic acid gel
- Hyaluronic acid+carrier (Active Comparator): hyaluronic acid gel application together with a carrier
  Interventions: Device: Hyaluronic acid gel + carrier
- Standard treatment (No Intervention): standard treatment (i.e., blood clot only)

INTERVENTIONS:
Device: Hyaluronic acid gel — After the local anesthesia is injected, alveolar curettage is performed, and the socket is rinsed with saline solution. Prior to wound closure, patients from the test group 1 will receive hyaluronic acid gel.
  Arms: Hyaluronic acid
Device: Hyaluronic acid gel + carrier — After the local anesthesia is injected, alveolar curettage is performed, and the socket is rinsed with saline solution. Prior to wound closure, patients from the test group 2 will receive hyaluronic acid gel together with a collagen carrier.
  Arms: Hyaluronic acid+carrier

SUMMARY:
Alveolar osteitis (AO; syn. dry socket) is one of the most frequent complications following tooth removal and it is defined as presence of severe postoperative pain in and around the extraction site, which increases in severity at any time between one and three days after extraction, accompanied by a partially or completely disintegrated blood cloth within the alveolar socket, with or without halitosis, and at the same time excluding any other cause for the pain (Blum 2002). To enhance standard treatment of AO, which consists of curettage of the dry socket, rinsing with saline solution, and inducing bleeding from the exposed alveolar bone walls, numerous products have been tested. One of them is hyaluronic acid (HY). The aim of the present study is to investigate the potential effect of HY gel application in the treatment of AO. Specifically, the application of HY only (HY test group; n = 20) or the combination of HY and an absorbable collagen sponge (HY+C test group; n = 20) will be compared to standard treatment (blood clot; control group, n=20). Clinical and patient related outcome parameters will be recorded for up to 14 days after treatment. A more stable blood clot and thus improved wound healing with faster pain reduction is expected through the use of HY.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years;
2. Untreated AO after extraction of a permanent tooth (excluding wisdom teeth);
3. Diagnosis of AO based on the criteria of Blum (Blum 2002)

   Exclusion Criteria:
4. Patients with chronic diseases and/or taking any medication, influencing hard and soft tissue healing;
5. Pregnancy;
6. History of hypersensitivity or allergy to HY;
7. Inability to attend follow-up appointments; Intake of preoperative antibiotics.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception by the patient | 2 weeks
  VAS- Visual analogue scale measured on a 10cm scale, where 0 represents no pain and 10 represents maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Dentistry, Medical University of Vienna, Vienna, Austria